CLINICAL TRIAL: NCT06406101
Title: Influence of CPR Surface Choice on Chest Compression Quality: A Randomized Manikin Study Comparing Bed and Floor Settings
Brief Title: CPR Surface Choice on Chest Compression Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Enrique Carrero, Director, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCBCPR_24147
Record Dates: First submitted 2024-05-03; First posted 2024-05-09 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Arrest; Simulation of Physical Illness
Keywords: Cardiopulmonary Resuscitation; Cardiac arrest; Simulation study; Chest Compressions
MeSH Terms: conditions — Heart Arrest | interventions — Floors and Floorcoverings; Beds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Floor (Experimental)
  Interventions: Other: Floor
- Bed (Active Comparator)
  Interventions: Other: Bed

INTERVENTIONS:
Other: Floor — Uninterrupted 2-minute chest compressions on a manikin that has been moved from the bed to the floor in a simulated scenario of out-of-hospital cardiac arrest
  Arms: Floor
Other: Bed — Uninterrupted 2-minute chest compressions on a manikin that is laying on bed in a simulated scenario of out-of-hospital cardiac arrest
  Arms: Bed

SUMMARY:
The objective of our randomized simulation study on mannequins with a population of Basic Life Support students is to compare the quality of chest compressions, taking depth as the main variable, in two simulated scenarios of out-of-hospital cardiac arrest on a bed: one where Cardiopulmonary Resuscitation is performed on the bed and another where the patient is transferred to the ground for Cardiopulmonary Resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Those individuals who sign the informed consent and do not meet exclusion criteria

Exclusion Criteria: Individuals with any limitation or contraindication for physical exercise:

* Arthritis
* Heart disease
* Advanced lung disease
* Severe physical disability
* Morbid obesity
* Chronic fatigue
* Pregnancy

Withdrawal Criteria:

* Those individuals who, due to limitations in physical exercise, do not reach 2 minutes of compressions
* Students who have not obtained the certificate of successfully completing the course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Compressions Mean Depth | On the day of the simulation
  Chest Compressions Mean Depth

SECONDARY OUTCOMES:
Time to first chest compression | On the day of the simulation
  The time it takes to initiate chest compressions.
Effectiveness of Chest Compressions | On the day of the simulation
  Global Punctuation of Chest Compressions in Skillreporter app.
Total number of chest compressions | On the day of the simulation
  Total number of chest compressions
Percentage of chest compressions whit correct depth (5-6cm) | On the day of the simulation
  Percentage of compressions whit correct depth (5-6cm)
Mean frequency of chest compressions | On the day of the simulation
  Mean frequency of chest compressions
Percentage of chest compressions with correct frequency | On the day of the simulation
  Percentage of chest compressions with correct frequency
Percentage of chest compressions with correct position of hands | On the day of the simulation
  Percentage of chest compressions with correct position of hands
Percentage of chest compressions with correct release | On the day of the simulation
  Percentage of chest compressions with correct release
Borg Scale for Fatigability | On the day of the simulation
  The scale includes a rating of 6 perceiving "no exertion at all" to 20 perceiving a "maximal exertion" of effort.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Capdevila, MD, Principal Investigator — Hospital Clinic Barcelona, Universitat de Barcelona
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided